CLINICAL TRIAL: NCT07008248
Title: Real-World Clinical Study for Malignant Tumor-Induced Cachexia
Status: Withdrawn | Type: Observational
Why Stopped: Company strategy adjustment
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Xuzhou Central Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: Megaxia RWS
Record Dates: First submitted 2025-05-26; First posted 2025-06-06 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2024-10

CONDITIONS: Clinical Characteristics and Treatment Outcomes of Malignant Tumor Cachexia; Multicenter Observational Study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective Cohort: This cohort focuses on patients who have already been diagnosed with cachexia before the initiation of this study. It involves the retrospective collection and analysis of clinical data.
- Prospective Cohort: This cohort includes patients who are diagnosed with cachexia after the start of this study. Data will be prospectively collected and analyzed during their subsequent diagnosis and treatment process.

SUMMARY:
This study is a non-interventional, multicenter observational study, aiming to assess the clinical characteristics and treatment outcomes of malignant tumor cachexia. The study is mainly divided into two cohorts:

Retrospective Cohort: This cohort focuses on patients who have already been diagnosed with cachexia before the initiation of this study. It involves the retrospective collection and analysis of clinical data.

Prospective Cohort: This cohort includes patients who are diagnosed with cachexia after the start of this study. Data will be prospectively collected and analyzed during their subsequent diagnosis and treatment process.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or older (including 18 years).
* Malignant tumor confirmed by histology or cytology (both malignant solid tumors and malignant hematologic tumors are eligible for enrollment).
* Meeting the Fearon diagnostic criteria for cachexia.
* Life expectancy of ≥2 months (for the prospective cohort only).
* Able to sign the informed consent form (waiver of informed consent for the retrospective cohort).

Exclusion Criteria:

Retrospective Cohort:

* Missing gender information.
* Missing date of birth or age information.
* Lack of any treatment or follow-up information after the date of meeting the diagnostic criteria for cachexia.

Prospective Cohort: (Patients with any of the following are not eligible for enrollment in this study)

* Patients who are unable to receive any treatment for any reason.
* Patients who cannot undergo at least one follow-up.
* Patients whom the investigator deems unsuitable for participation in this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cachexia patients with malignant tumors
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2024-10-15 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
The value of weight increase compared to the baseline | through the observation period，an average of 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Xuzhou Central Hospital, Xuzhou Clinical School of Xuzhou Medical University, Xuzhou, Jiangsu, China